CLINICAL TRIAL: NCT06057324
Title: Switching Mediterranean Consumers to Mediterranean Sustainable Healthy Dietary Patterns by Combining Digital Interactive Tools with Targeted Educational Material and Sustainable Snacks
Brief Title: Switching Mediterranean Consumers to Mediterranean Sustainable Healthy Dietary Patterns
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: Centre de Recerca en Economia i Desenvolupament Agroalimentari-UPC-IRTA (CREDA) (Unknown); Unité Mixte de Recherche en Nutrition et Alimentation, Université Ibn Tofail (CNESTEN) (Unknown); Uludag University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SWITCHtoHEALTHY; 2133 (Other Grant/Funding Number: European Union Funding for Research and Innovation - HORIZON 2020)
Record Dates: First submitted 2023-08-04; First posted 2023-09-28 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Healthy Subjects; Behavior, Health; Family
Keywords: Mediterranean Diet; Adherence; Family; Nutritional intervention; Sustainability; Educational Activities; Healthy Food Choice; Digital Technology; Healthy food
MeSH Terms: conditions — Health Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Multicentre, parallel, randomized, single-blind and controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, the participating families and researchers cannot be blinded to the intervention, although the researchers who will perform the data analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multi-component intervention groups (Experimental): Multi-component intervention with non-invasive approaches:
  -Digital interactive tools (AI-based Apps): They will consist of a combination of two Artificial Intelligence (AI) Apps that will be used by parents to empower them in their daily dietary choices for children's dietary plan.
  - Educational materials (Mediterranean-based diet toolkit) and activities: The toolkit will include a set of specific games and activities for kids designed to facilitate the ''learning through playing'' approach improving their understanding of different nutrition themes. The educational activities will be co-designed and carried out by adolescents outside of school hours.
  - Healthy plant-based snacks: They will be adapted to children's nutritional requirements and to be consumed in-between time on a daily basis. Based on local and traditional products for each country including vegetables, fruits, legumes, seeds and nuts as main ingredients.
  Interventions: Device: AI-based Apps; Behavioral: Mediterranean-based diet toolkit and activities; Other: Healthy plant-based snacks; Other: AI-based Apps + Mediterranean-based diet toolkit and activities; Other: AI-based Apps + Healthy plant-based snacks; Other: Mediterranean-based diet toolkit and activities + Healthy plant-based snacks; Other: AI-based Apps + Mediterranean-based diet toolkit and activities + Healthy plant-based snacks
- Control group (No Intervention): Families which will not follow any intervention; they will receive basic Mediterranean guidelines for parents and their children.

INTERVENTIONS:
Device: AI-based Apps — Families which will use the digital interactive tools to empower parents in their daily dietary choices.
  Arms: Multi-component intervention groups
Behavioral: Mediterranean-based diet toolkit and activities — Families which will receive educational materials and adolescents will perform educational activities.
  Arms: Multi-component intervention groups
Other: Healthy plant-based snacks — Families in which children will include the snacks in their diet.
  Arms: Multi-component intervention groups
Other: AI-based Apps + Mediterranean-based diet toolkit and activities — Families which will use the digital interactive tools and receive educational material, and adolescents will perform educational activities.
  Arms: Multi-component intervention groups
Other: AI-based Apps + Healthy plant-based snacks — Families which will use the digital interactive tools and children will include the snacks in their diet.
  Arms: Multi-component intervention groups
Other: Mediterranean-based diet toolkit and activities + Healthy plant-based snacks — Families which will receive educational material, adolescents will perform educational activities, and children will include the snacks in their diet.
  Arms: Multi-component intervention groups
Other: AI-based Apps + Mediterranean-based diet toolkit and activities + Healthy plant-based snacks — Families which will use the digital interactive tools and will receive educational material, children will include the snacks in their diet, and adolescents will perform educational activities.
  Arms: Multi-component intervention groups

SUMMARY:
The population from Mediterranean countries is abandoning the Mediterranean diet (MD) traditional dietary and lifestyle pattern moving to unhealthier habits because of profound cultural and socio-economic driven lifestyle changes. Families, particularly parents, are responsible for structuring children's early experiences with food and eating as well as for transmitting knowledge of the MD. Educational family approaches can not only lead to more solid food literacy and healthy habits for children in the family but can also improve dietary profiles for adults, thus preventing future health-related problems. There is a lack of adequate study protocol for inducing a positive dietary, environmental and lifestyle behaviour in the family setting. SWITCHtoHEALTHY study aims to evaluate the effects of a multi-component nutritional intervention deployed at family level on the adherence to the MD pattern in families from three Mediterranean countries.

A parallel, randomized, single blind controlled multicentric nutritional intervention study will be conducted in 480 families with children and adolescents among 3-17 years from Spain, Morocco, and Turkey over 13 months. Specifically, 160 families per country will be enrolled in a multi-component intervention and allocated to use digital interactive tools, hands-on educational materials and activities for adolescents, easy-to-eat healthy plant-based snacks for children, or a combination of two or three of the components. There will also be a control group that will receive general advice on healthy eating. The intervention study is scheduled to begin in November 2023.

Through the digital tools the parents will use an interactive App through which they will receive personalized weekly meal plans while the engagement of all the family will be prompted by using a life simulation game. A set of activities for adolescents based on a learning-through-play approach to be carried out within the family and at school will be developed by adolescents and voluntary schoolteachers through co-creation sessions. The innovative and sustainable plant-based snacks will be produced by local food companies and introduced in the children dietary plan as healthy alternatives for between meals. By using a full-factorial design, the independent and combined effects of each intervention component will be tested by comparing the 7 intervention groups with the control group.

DETAILED DESCRIPTION:
The main outcome will be adherence to the MD assessed through MEDAS and KIDMED validated questionnaires in parents and children respectively. The effectiveness of the multi-component intervention will be evaluated by comparing the MEDAS and KIDMED scores between the control and intervention groups at baseline and at the end of the intervention.The secondary outcomes will include a set of anthropometrical, lifestyle, dietary and socio-economic indicators measured in all family members.

Standardized protocols will be used for the collection of data in the three countries. All data will be collected and evaluated by professional researchers and registered by researchers or study participants in a web platform. Lifestyle, diet, and socio-economic indicators will be self-reported by means of adapted online questionnaires for parent, adolescent, and child.

The study will be carried out in 2 phases:

* Phase 1 (month 0 to month 9): the families will be included in the study, they will be assigned to the different intervention groups, and consumption patterns and lifestyle, diet, and socioeconomic indicators will be evaluated through specific questionnaires. In addition, the different educational materials, activities, digital interactive tools and healthy snacks will be developed prior to the start of the intervention study.
* Phase 2 (month 10 to month 13): The intervention study will be deployed at family level. Each family will receive the educational materials, digital interactive tools and snacks developed in Phase 1 as assigned. In addition, anthropometric, lifestyle, dietary and socioeconomic indicators will be evaluated through questionnaires.

Three visits will be performed along the study, including one pre-assessment at the beginning of Phase 1 (baseline, month 0), one visit at the beginning of Phase 2 (month 11) and one visit at the end of Phase 2 (month 13).

The impact of the intervention on dietary factors, including MD adherence, diet quality, food intake and MD lifestyle habits, physical activity, and classical anthropometrical parameters, will be assessed in Phase 2 in a 3-month period. However, consumption behaviour and environmental and economic factors will be measured at the baseline (Phase 1) and at the end (Phase 2). The baseline point (month 0) is necessary to assess the aforementioned factors over the course of a year.

ELIGIBILITY:
Inclusion Criteria:

* Families from any socioeconomic status with at least one child less than 12 years and one adolescent older than or equal to 12 years (overall age range 3 - 17 years) and that live together.
* Signed informed consent (parents will sign on their own behalf and of the child under 12 years of age and the adolescent. The adolescent must also sign themselves).
* To have a mobile phone, tablet, or computer with internet access.

Exclusion Criteria:

* Having allergies or food intolerances to any of the snack ingredients: fruit, vegetables, legumes, cereals, seeds, nuts (only for children under 12 years).
* Dislike any of the snacks (only for children under 12 years).
* Mediterranean Diet Adherence Score (MEDAS) among 8-14 or KIDMED score among 8-12, which is a food pattern already highly concordant with the Mediterranean Diet.
* Following a vegan diet any of the family members.
* Following a prescribed long-term and strict diet for any reason, including diets for weight loss and diets for chronic metabolic or autoimmune disorders such as type 1 diabetes, celiac disease, inflammatory bowel disease or rheumatoid arthritis (any of the family members).
* Participate in or have participated in a clinical trial or nutritional intervention study in the last 30 days prior to inclusion in the study.
* No or limited access to the Internet.
* Being unable to follow the study guidelines.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in adherence to the Mediterranean Diet | Phase 2 (month 10 to month 13)
  The main outcome will be adherence to the MD measured through MEDAS questionnaire score in parents. The effectiveness of the multi-component intervention will be evaluated by comparing the MEDAS score between the control and intervention groups during the intervention period (Phase 2).
  The MEDAS score is an extension of a 9-point score developed in the Prevention with Mediterranean Diet (PREDIMED) trial. A score of 14 points means maximum adherence to the Mediterranean Diet while a score below 7 points means low adherence.
Change in adherence to the Mediterranean Diet | Phase 2 (month 10 to month 13)
  The main outcome will be adherence to the MD measured through KIDMED questionnaire score in children. The effectiveness of the multi-component intervention will be evaluated by comparing the KIDMED score between the control and intervention groups during the intervention period (Phase 2).
  The KIDMED score ranges from 0 to 12 points, so a score greater than or equal to 8 points means optimal Mediterranean Diet adherence while a score below or equal to 3 points means very low-quality diet, and between 4 and 7 points means that need to improve the eating pattern to fit the Mediterranean pattern.

SECONDARY OUTCOMES:
Change in Body Mass Index values | Phase 2 (month 10 to month 13)
  BMI will be assessed by weight (kg) / height (m2) and using a body composition analyzer (Tanita). BMI values will be compared between control and intervention groups. Measured in all family members.
Change in waist circumference values | Phase 2 (month 10 to month 13)
  Waist circumference (cm) will be measured at the umbilicus level using an anthropometric steel measuring tape. The obtained values will be compared between control and intervention groups. Measured in all family members.
Change in blood pressure values | Phase 2 (month 10 to month 13)
  Systolic blood pressure and Diastolic blood pressure values (mmHg) will be monitored by using an automatic sphygmomanometer. The obtained results will be compared between control and intervention groups. Measured in all family members.
Change in resting heart rate values | Phase 2 (month 10 to month 13)
  Resting heart rate values (bpm) will be monitored by using an automatic sphygmomanometer. The obtained results will be compared between control and intervention groups. Measured in all family members.
Sociodemographic and socioeconomic data | Phase 1 (baseline)
  Measured in parents and adolescents by an adapted questionnaire which will collect information regarding age, gender, household members, marital status, income, level of education and employment status.
Social factors data | Phase 1 (baseline)
  Measured in parents, adolescents, and children over 8 years by an adapted questionnaire which will collect information regarding work flexibility and satisfaction, work-life balance, lifestyle, time spent with children, family decision making, and task responsibility.
Change in physical activity levels | Phase 2 (month 10 to month 13)
  Physical activity level will be measured by using the Physical Activity Questionnaires PAQ-C for children over 8 years. It consists of a 10-item validated scale. The resulting score ranges from 1 to 5. A score of 1 indicates low physical activity, whereas a score of 5 indicates high physical activity. The obtained scores will be compared between control and intervention groups.
Change in physical activity levels | Phase 2 (month 10 to month 13)
  Physical activity level will be measured by using the International Physical Activity Questionnaire (IPAQ) for adults (parents). It consists of a 7-item short form with open-ended questions surrounding individuals' last 7-day recall of physical activity. Results are reported as categories (low activity levels, moderate activity levels or high activity levels). The obtained results will be compared between control and intervention groups.
Change in quality of life | Phase 2 (month 10 to month 13)
  Quality of life will be measured by using the 5-level EQ-5D-5L scale (EuroQol Group) for adults (parents). The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The subject is asked to indicate his/her health state in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state. The obtained scores will be compared between control and intervention groups.
Change in quality of life | Phase 2 (month 10 to month 13)
  Quality of life will be measured by using the KIDSCREEN questionnaire for adolescents and children over 8 years. This scale measures 10 health-related quality of life dimensions: Physical- (5 items), Psychological Well-being (6 items), Moods and Emotions (7 items), Self-Perception (5 items), Autonomy (5 items), Parent Relations and Home Life (6 items), Social Support and Peers (6 items), School Environment (6 items), Social Acceptance (Bullying) (3 items), Financial Resources (3 items). The obtained scores will be compared between control and intervention groups.
Change in nutritional knowledge | Phase 2 (month 10 to month 13)
  Knowledge about food and nutrition will be measured using a short consumer-oriented nutrition knowledge questionnaire for adults. The questionnaire consists of a scale of 20 items where correct responses are scored as one, while incorrect responses, don't know-answers or blanks are scored as zero. The obtained final scores will be compared between control and intervention groups.
Change in nutritional knowledge | Phase 2 (month 10 to month 13)
  Knowledge about food and nutrition will be measured using the HELENA (Healthy Lifestyle in Europe by Nutrition in Adolescence) study questionnaire for adolescents. The questionnaire includes a total of 23 multiple-choice questions that can be categorized into specific subscales regarding knowledge of concepts (e.g. subscales 'Energy Intake and Energy Metabolism' or 'Physical Activity'), instrumental knowledge (e.g. subscale 'Nutrient Contents') and knowledge of causal relationships (e.g. subscales 'Sweeteners' or 'Oral Health'). Each question offers three possible answers (only one correct) and the 'don't know' category. Correct answers are scored as 1 and incorrect answers are scored as 0. Finally, the individual scores are summed up and calculated as a percentage of the total. The obtained final scores will be compared between control and intervention groups.
Change in the health factor | Phase 1 (month 0 to month 9) and Phase 2 (month 10 to month 13)
  The health factor will be assessed by the General Health Questionnaire (GHQ). This questionnaire will ask different aspects related to health and healthy lifestyle such as sleeping habits, hospitalization, or prescribed medications. The obtained results will be compared between control and intervention groups. Measured in all family members.
Change in Mediterranean Diet lifestyle habits | Phase 1 (month 0 to month 9) and Phase 2 (month 10 to month 13)
  Measured in parents by the Mediterranean Lifestyle index (MEDLIFE), which will capture adherence to an overall Mediterranean healthy lifestyle. It consists of a 28-item questionnaire categorized into three blocks: (1) Mediterranean food consumption (15 items); (2) Mediterranean dietary habits (7 items); (3) Physical Activity, rest, social habits and conviviality (6 items). Each item is scored as 0 for not meeting the cutoff established for the item or 1 for meeting it, so that the complete MEDLIFE ranges from 0 to 28, with a higher value indicative of greater adherence to Mediterranean lifestyle. The obtained results will be compared between control and intervention groups.
Change in diet quality | Phase 1 (month 0 to month 9) and Phase 2 (month 10 to month 13)
  Diet quality will be measured by using the Healthy Diet Index (HDI) for adults. It consists of seven weighted domains (meal pattern, grains, fruit and vegetables, fats, fish and meat, dairy, snacks, and treats). Within each domain, increasing points indicate a more healthy diet. The maximum total HDI is set at 100 points. The obtained results will be compared between control and intervention groups.
Change in diet quality | Phase 1 (month 0 to month 9) and Phase 2 (month 10 to month 13)
  Diet quality will be measured by using the KIDMED questionnaire for adolescent and children. The KIDMED score ranges from 0 to 12 points, so a score greater than or equal to 8 points means optimal diet quality while a score below or equal to 3 points means very low-quality diet, and between 4 and 7 points means that need to improve the eating pattern. The obtained score will be compared between control and intervention groups.
Change in attitudes and beliefs in relation to food | Phase 1 (month 0 to month 9) and Phase 2 (month 10 to month 13)
  Measured by an adapted questionnaire for parents. This questionnaire measures how the household income, parents' time spent with children, and parents' work experiences affect children's energy and fat intake and obesity-related outcomes. The obtained results will be compared between control and intervention groups.
Change in consumption behavior | Phase 1 (month 0 to month 9) and Phase 2 (month 10 to month 13)
  The consumption patterns will be assessed by means of family weekly food purchases, food intakes and food waste. The food purchases will be monitored by family unit using shopping tickets collected for 1 week. The food intake will be measured in all family by a 7-day semi-weighted food record. The food waste will be calculated as the difference between families food purchases and consumption considering the initial and final food inventories. Food storage sheets will be used to estimate the balance between food purchased and stored at home.
Change in environmental impact | Phase 1 (month 0 to month 9) and Phase 2 (month 10 to month 13)
  The environmental impact of food consumption will be assessed of the overall study and the intervention. The consumption quantities will be converted into kg of CO2 emission, land use and water footprint using existing tables in the literature on the environmental impacts of different food groups.
Change in economic impact | Phase 1 (month 0 to month 9) and Phase 2 (month 10 to month 13)
  The economic impact of the overall study and the intervention will be estimated using the family shopping tickets. We will evaluate whether the interventions lead to any change in family food expenditures.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari Palou, PhD, Principal Investigator — Fundació Eurecat
Locations (1):
- Eurecat, Technological Center of Catalonia, Nutrition and Health Unit, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alonso-Dominguez R, Garcia-Ortiz L, Patino-Alonso MC, Sanchez-Aguadero N, Gomez-Marcos MA, Recio-Rodriguez JI. Effectiveness of A Multifactorial Intervention in Increasing Adherence to the Mediterranean Diet among Patients with Diabetes Mellitus Type 2: A Controlled and Randomized Study (EMID Study). Nutrients. 2019 Jan 14;11(1):162. doi: 10.3390/nu11010162. PMID 30646500
- [Background] Sichert-Hellert W, Beghin L, De Henauw S, Grammatikaki E, Hallstrom L, Manios Y, Mesana MI, Molnar D, Dietrich S, Piccinelli R, Plada M, Sjostrom M, Moreno LA, Kersting M; HELENA Study Group. Nutritional knowledge in European adolescents: results from the HELENA (Healthy Lifestyle in Europe by Nutrition in Adolescence) study. Public Health Nutr. 2011 Dec;14(12):2083-91. doi: 10.1017/S1368980011001352. Epub 2011 Aug 2. PMID 21810282
- [Background] Dickson-Spillmann M, Siegrist M, Keller C. Development and validation of a short, consumer-oriented nutrition knowledge questionnaire. Appetite. 2011 Jun;56(3):617-20. doi: 10.1016/j.appet.2011.01.034. Epub 2011 Feb 15. PMID 21310201
- [Background] Ravens-Sieberer U, Gosch A, Abel T, Auquier P, Bellach BM, Bruil J, Dur W, Power M, Rajmil L; European KIDSCREEN Group. Quality of life in children and adolescents: a European public health perspective. Soz Praventivmed. 2001;46(5):294-302. doi: 10.1007/BF01321080. PMID 11759336
- [Background] Sotos-Prieto M, Santos-Beneit G, Bodega P, Pocock S, Mattei J, Penalvo JL. VALIDATION OF A QUESTIONNAIRE TO MEASURE OVERALL MEDITERRANEAN LIFESTYLE HABITS FOR RESEARCH APPLICATION: THE MEDITERRANEAN LIFESTYLE INDEX (MEDLIFE). Nutr Hosp. 2015 Sep 1;32(3):1153-63. doi: 10.3305/nh.2015.32.3.9387. PMID 26319833
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Rodriguez-Rodriguez F, Galvez-Fernandez P, Huertas-Delgado FJ, Aranda-Balboa MJ, Saucedo-Araujo RG, Herrador-Colmenero M. Parent's sociodemographic factors, physical activity and active commuting are predictors of independent mobility to school. Int J Health Geogr. 2021 Jun 6;20(1):26. doi: 10.1186/s12942-021-00280-2. PMID 34090437
- [Background] Serra-Majem L, Ribas L, Ngo J, Ortega RM, Garcia A, Perez-Rodrigo C, Aranceta J. Food, youth and the Mediterranean diet in Spain. Development of KIDMED, Mediterranean Diet Quality Index in children and adolescents. Public Health Nutr. 2004 Oct;7(7):931-5. doi: 10.1079/phn2004556. PMID 15482620
- [Background] Quintana-Navarro GM, Alcala-Diaz JF, Lopez-Moreno J, Perez-Corral I, Leon-Acuna A, Torres-Pena JD, Rangel-Zuniga OA, Arenas de Larriva AP, Corina A, Camargo A, Yubero-Serrano EM, Rodriguez-Cantalejo F, Garcia-Rios A, Luque RM, Ordovas JM, Perez-Martinez P, Lopez-Miranda J, Delgado-Lista J. Long-term dietary adherence and changes in dietary intake in coronary patients after intervention with a Mediterranean diet or a low-fat diet: the CORDIOPREV randomized trial. Eur J Nutr. 2020 Aug;59(5):2099-2110. doi: 10.1007/s00394-019-02059-5. Epub 2019 Jul 24. PMID 31342228
- [Background] Martinez-Gonzalez MA, Garcia-Arellano A, Toledo E, Salas-Salvado J, Buil-Cosiales P, Corella D, Covas MI, Schroder H, Aros F, Gomez-Gracia E, Fiol M, Ruiz-Gutierrez V, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Munoz MA, Warnberg J, Ros E, Estruch R; PREDIMED Study Investigators. A 14-item Mediterranean diet assessment tool and obesity indexes among high-risk subjects: the PREDIMED trial. PLoS One. 2012;7(8):e43134. doi: 10.1371/journal.pone.0043134. Epub 2012 Aug 14. PMID 22905215
- [Background] Leblanc V, Begin C, Hudon AM, Royer MM, Corneau L, Dodin S, Lemieux S. Effects of a nutritional intervention program based on the self-determination theory and promoting the Mediterranean diet. Health Psychol Open. 2016 Jan 3;3(1):2055102915622094. doi: 10.1177/2055102915622094. eCollection 2016 Jan. PMID 28070382
- [Background] Chakraborty B, Collins LM, Strecher VJ, Murphy SA. Developing multicomponent interventions using fractional factorial designs. Stat Med. 2009 Sep 20;28(21):2687-708. doi: 10.1002/sim.3643. PMID 19575485
- [Background] Harris JL, Romo-Palafox MJ, Gershman H, Kagan I, Duffy V. Healthy Snacks and Drinks for Toddlers: A Qualitative Study of Caregivers' Understanding of Expert Recommendations and Perceived Barriers to Adherence. Nutrients. 2023 Feb 17;15(4):1006. doi: 10.3390/nu15041006. PMID 36839364
- [Background] Black AP, D'Onise K, McDermott R, Vally H, O'Dea K. How effective are family-based and institutional nutrition interventions in improving children's diet and health? A systematic review. BMC Public Health. 2017 Oct 17;17(1):818. doi: 10.1186/s12889-017-4795-5. PMID 29041899
- [Background] Bibiloni MDM, Gallardo-Alfaro L, Gomez SF, Warnberg J, Oses-Recalde M, Gonzalez-Gross M, Gusi N, Aznar S, Marin-Cascales E, Gonzalez-Valeiro MA, Serra-Majem L, Terrados N, Segu M, Lassale C, Homs C, Benavente-Marin JC, Labayen I, Zapico AG, Sanchez-Gomez J, Jimenez-Zazo F, Alcaraz PE, Sevilla-Sanchez M, Herrera-Ramos E, Pulgar S, Sistac C, Schroder H, Bouzas C, Tur JA. Determinants of Adherence to the Mediterranean Diet in Spanish Children and Adolescents: The PASOS Study. Nutrients. 2022 Feb 9;14(4):738. doi: 10.3390/nu14040738. PMID 35215388
- [Background] Iaccarino Idelson P, Scalfi L, Valerio G. Adherence to the Mediterranean Diet in children and adolescents: A systematic review. Nutr Metab Cardiovasc Dis. 2017 Apr;27(4):283-299. doi: 10.1016/j.numecd.2017.01.002. Epub 2017 Jan 12. PMID 28254269
- [Background] Nasreddine L, Ayoub JJ, Al Jawaldeh A. Review of the nutrition situation in the Eastern Mediterranean Region. East Mediterr Health J. 2018 Apr 5;24(1):77-91. PMID 29658624
- [Background] Dai H, Alsalhe TA, Chalghaf N, Ricco M, Bragazzi NL, Wu J. The global burden of disease attributable to high body mass index in 195 countries and territories, 1990-2017: An analysis of the Global Burden of Disease Study. PLoS Med. 2020 Jul 28;17(7):e1003198. doi: 10.1371/journal.pmed.1003198. eCollection 2020 Jul. PMID 32722671
- [Background] GBD 2017 Diet Collaborators. Health effects of dietary risks in 195 countries, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 May 11;393(10184):1958-1972. doi: 10.1016/S0140-6736(19)30041-8. Epub 2019 Apr 4. PMID 30954305
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med. 2013 Apr 4;368(14):1279-90. doi: 10.1056/NEJMoa1200303. Epub 2013 Feb 25. PMID 23432189 (Retraction: PMID 29897867 N Engl J Med. 2018 Jun 21;378(25):2441-2442)
- [Background] Tuttolomondo A, Simonetta I, Daidone M, Mogavero A, Ortello A, Pinto A. Metabolic and Vascular Effect of the Mediterranean Diet. Int J Mol Sci. 2019 Sep 23;20(19):4716. doi: 10.3390/ijms20194716. PMID 31547615
- [Derived] Calderon-Perez L, Domingo A, Bas JMD, Gutierrez B, Crescenti A, Rahmani D, Sarroca A, Gil JM, Goumeida K, Zhang Jin T, Guldas M, Demir CE, Hamdouchi AE, Gymnopoulos LP, Dimitropoulos K, Degli Innocenti P, Rosi A, Scazzina F, Petri E, Urtasun L, Salvio G, Feld M, Boque N. Switching Mediterranean Consumers to Mediterranean Sustainable Healthy Dietary Patterns (SWITCHtoHEALTHY): Study Protocol of a Multicentric and Multi-Cultural Family-Based Nutritional Intervention Study. Nutrients. 2024 Nov 18;16(22):3938. doi: 10.3390/nu16223938. PMID 39599724